CLINICAL TRIAL: NCT06503783
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of BL-M17D1 in Patients With Locally Advanced or Metastatic HER2 Positive/Negative Breast Cancer and Other Solid Tumors
Brief Title: A Study of BL-M17D1 in Patients With Locally Advanced or Metastatic HER2 Positive/Negative Breast Cancer and Other Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-M17D1-101
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Solid Tumor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-M17D1 (Experimental): Participants receive BL-M17D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M17D1

INTERVENTIONS:
Drug: BL-M17D1 — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This study is an open, multicenter, dose-escalation and expansion-enrollment nonrandomized phase I clinical study to evaluate the safety, tolerability, pharmacokinetic characteristics and preliminary efficacy of BL-M17D1 in patients with locally advanced or metastatic HER2 positive/negative breast cancer and other solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Gender is not limited;
3. Age: ≥18 years old and ≤75 years old (stage Ia); ≥18 years old (stage Ib);
4. Expected survival time ≥3 months;
5. Patients with locally advanced or metastatic HER2-positive/negative breast cancer and other solid tumors;
6. Agree to provide archival tumor tissue samples or fresh tissue samples of primary or metastatic lesions within 3 years;
7. Must have at least one extracranial measurable lesion that meets the RECIST v1.1 definition;
8. ECOG 0 or 1;
9. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. No blood transfusion is allowed within 14 days before the first use of the study drug, and no cell growth factor is allowed. The organ function level must meet the requirements;
12. Coagulation function: international normalized ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5ULN;
13. For premenopausal women of childbearing potential, a pregnancy test must be performed within 7 days before the initiation of treatment, serum pregnancy must be negative, and the patient must not be lactating; All enrolled patients (male or female) were advised to use adequate barrier contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Chemotherapy, biological therapy and other anti-tumor therapies have been used within 4 weeks or 5 half-lives before the first dose; Mitomycin and nitrosoureas were administered within 6 weeks before the first dose; Oral drugs such as fluorouracil;
2. History of severe heart disease;
3. Prolonged QT interval, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
4. Active autoimmune and inflammatory diseases;
5. Other malignancies diagnosed within 5 years before the first dose;
6. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening; Infusion-related thrombosis was excluded;
7. Hypertension poorly controlled by two antihypertensive drugs (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg);
8. A history of ILD requiring steroid therapy, or current ILD or radiation pneumonitis of grade ≥1 according to the RTOG/EORTC definition, or a suspicion of such disease;
9. Patients with poor glycemic control;
10. Complicated with pulmonary diseases leading to clinically severe respiratory function impairment;
11. Patients with primary central nervous system tumors or CNS metastases after failure of local treatment;
12. Patients with a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or to any of BL-M17D1's excipients;
13. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation;
14. Prior anthracycline therapy with more than the protocol-specified cumulative dose of an anthracycline;
15. Human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection or active hepatitis C virus infection;
16. Active infection requiring systemic therapy with a serious infection within 4 weeks prior to informed consent; There were indications of pulmonary infection or active pulmonary inflammation within 2 weeks before informed consent;
17. Patients with massive or symptomatic effusions, or poorly controlled effusions;
18. Had participated in another clinical trial within 4 weeks before the first dose;
19. Pregnant or lactating women;
20. Patients with superior vena cava syndrome should not be rehydrated;
21. A history of severe neurological or psychiatric illness;
22. Severe unhealed wounds, ulcers, or fractures within 4 weeks before signing the informed consent;
23. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
24. History of intestinal obstruction, inflammatory bowel disease or extensive bowel resection or presence of Crohn's disease, ulcerative colitis or chronic diarrhea;
25. Who are scheduled to receive live vaccine or who receive the vaccine within 28 days before the first dose;
26. The investigators did not consider it appropriate to apply other conditions for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose limiting toxicity (DLT) | Up to 21 days after the first dose
  DLTs are assessed according to NCI-CTCAE v5.0 during the first cycle and defined as occurrence of any of the toxicities in DLT definition if judged by the investigator to be possibly, probably or definitely related to study drug administration.
Phase Ia: Maximum tolerated dose (MTD) | Up to 21 days after the first dose
  MTD is defined as the highest dose level at which no more than 1 in 6 participants experienced a DLT during the first cycle .
Phase Ib: Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-M17D1.

SECONDARY OUTCOMES:
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M17D1 . The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M17D1.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-M17D1 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of BL-M17D1 will be investigated.
T1/2 | Up to approximately 24 months
  Half-life (T1/2) of BL-M17D1 will be investigated.
AUC0-t | Up to approximately 24 months
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration.
CL (Clearance) | Up to approximately 24 months
  CL in the serum of BL-M17D1 per unit of time will be investigated.
Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of BL-M17D1 prior to the next dose will be administered.
ADA (anti-drug antibody) | Up to approximately 24 months
  Frequency of anti-BL-M17D1 antibody (ADA) will be investigated.
Phase Ib: Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Phase Ib: Disease Control Rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Phase Ib: Duration of Response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality